CLINICAL TRIAL: NCT00233129
Title: Improving Executive Functions After TBI: A Randomized Clinical Trial of the "Executive Plus" Program
Brief Title: Improving Executive Functions After Traumatic Brain Injury (TBI): A Clinical Trial of the "Executive Plus" Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO# 04-0782; #H133B040033
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Traumatic Brain Injury
Keywords: Day treatment; executive function; problem solving; attention; participation; TBI; brain injury; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (Active Comparator): cognitive rehabilitation day treatment program
  Interventions: Other: cognitive rehabilitation day treatment program
- Top-Down (Experimental): cognitive rehabilitation day treatment program that incorporates systematic "top down" treatment of executive function deficits (problem solving and emotional regulation training), systematic treatment of attention deficits, and modular, contextual and embedded approaches to treatment.
  Interventions: Behavioral: Top Down

INTERVENTIONS:
Behavioral: Top Down — Six months
  Other Names: Executive Plus Day Treatment Program
  Arms: Top-Down
Other: cognitive rehabilitation day treatment program — six months
  Arms: Standard Treatment

SUMMARY:
This is a randomized clinical trial which compares a standard day treatment program for individuals with TBI with the "Executive Plus" program; the latter emphasizes training of attention, emotional self-regulation and problem solving. The goal of the Executive Plus program is to maximize executive functioning, as well as the long-term outcomes of community participation and satisfaction with daily life.

DETAILED DESCRIPTION:
This is a randomized clinical trial comparing two approaches to post-TBI comprehensive day treatment. Executive Plus offers systematic treatment of post-TBI executive function deficits, through a focus on problem solving and emotional self-regulation, as well as systematic treatment of post-TBI attention deficits. It relies on modular, contextual, and embedded approaches to treatment. It will be compared to Mount Sinai's currently operating day treatment program. The 26-week programs will run concurrently and potential participants will be randomly assigned to Executive Plus or the standard program, using rolling admissions. Program staffs will be separate. Outcomes will be assessed using measures that focus on functioning within cognitive domains, across domains and in everyday life, and that assess long-term outcomes. Detailed manuals will be developed to guide the implementation of each program's operation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Having a TBI as a result of a blow to the head followed by a loss of consciousness or period of being dazed and confused or a period of post traumatic amnesia or clinical signs of altered neurological function; this information must be medically documented (e.g., emergency medical record, hospital record, neuroradiological report, or neurological exam or record of physician's visit within 24 hours of injury).
* At least three months post-injury
* English-speaking (treatment sessions will be conducted in English)
* Reporting executive dysfunction (by self or family)
* Willing and able to participate in and travel to the program daily for six months
* Oriented to time, place and person
* Having a full-scale intelligence quotient (IQ) of at least 75
* Having a score on the Galveston Orientation and Amnesia Test of 75 or more
* Having communication skills adequate to participate in groups
* Having at least a sixth-grade reading level (for testing and use of written materials)
* Willing to complete questionnaires and interviews about mood, thinking skills, participation and the like
* Agree to participate, i.e., completion of informed consent and Health Insurance Portability and Accountability Act (HIPAA) documents

Exclusion Criteria:

* Active substance abuse
* Active psychosis
* Active suicidality
* Disruptive or violent behavior to self or others
* Current cognitive rehabilitation (this does not include psychotherapy)
* No impairment on the Frontal Systems Behavior Scale (FRSBE) or Wisconsin Card Sorting Test (WCST)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Cognitive function | At baseline
Cognitive function | 5 weeks into treatment
Cognitive function | At treatment end (6 months after baseline)
Cognitive function | 6 months after completing treatment
Cognitive function | 12 months after completing treatment

SECONDARY OUTCOMES:
Memory | At baseline
Memory | 5 weeks into treatment
Memory | At treatment end (6 months after baseline)
Memory | 6 months after completing treatment
Memory | 12 months after completing treatment
Learning | At baseline
Learning | 5 weeks into treatment
Learning | At treatment end (6 months after baseline)
Learning | 6 months after completing treatment
Learning | 12 months after completing treatment
Participation | At baseline
Participation | 5 weeks into treatment
Participation | At treatment end (6 months after baseline)
Participation | 6 months after completing treatment
Participation | 12 months after completing treatment
Affective distress | At baseline
Affective distress | 5 weeks into treatment
Affective distress | At treatment end (6 months after baseline)
Affective distress | 6 months after completing treatment
Affective distress | 12 months after completing treatment
Life satisfaction and self-efficacy | At baseline
Life satisfaction and self-efficacy | 5 weeks into treatment
Life satisfaction and self-efficacy | At treatment end (6 months after baseline)
Life satisfaction and self-efficacy | 6 months after completing treatment
Life satisfaction and self-efficacy | 12 months after completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wayne A Gordon, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States